CLINICAL TRIAL: NCT05668403
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profiles and Preliminary Efficacy of Subcutaneous Injection of Recombinant Humanized Anti-CD20 Monoclonal Antibody in the Treatment of Primary Membranous Nephropathy
Brief Title: A Phase I Clinical Study of Recombinant Humanized Anti-CD20(B-lymphocyte Antigen CD20) Monoclonal Antibody Subcutaneous Injection in the Treatment of Primary Membranous Nephropathy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiaolian Drug Research and Development Co., Ltd (Industry)
Collaborators: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: B007-102
Record Dates: First submitted 2022-12-12; First posted 2022-12-29 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Primary Membranous Nephropathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- B007:350mg (Experimental): B007:350mg Subcutaneous injection was administered on days 1 and 15
  B007 matched Placebo Subcutaneous injection was administered on days 1 and 15
  Interventions: Drug: B007
- B007:700mg (Experimental): B007: 700mg Subcutaneous injection was administered on days 1 and 15
  B007 matched Placebo Subcutaneous injection was administered on days 1 and 15
  Interventions: Drug: B007
- B007:1000mg (Experimental): B007: 1000mg Subcutaneous injection was administered on days 1 and 15
  B007 matched Placebo Subcutaneous injection was administered on days 1 and 15
  Interventions: Drug: B007

INTERVENTIONS:
Drug: B007 — Drug: B007 injection Drug: Placebo injection
  Arms: B007:350mg
Drug: B007 — Drug: B007 injection Drug: Placebo injection
  Arms: B007:700mg
Drug: B007 — Drug: B007 injection Drug: Placebo injection
  Arms: B007:1000mg

SUMMARY:
This Phase I Clinical Study assessed the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profiles and Preliminary Efficacy of Subcutaneous Injection of Recombinant Humanized Anti-CD20 Monoclonal Antibody in the Treatment of Primary Membranous Nephropathy

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have fully understood this study and voluntarily signed the informed consent form;
2. Male or female subjects, aged between 18 and 75 years;
3. Subjects with primary membranous nephropathy pathologically confirmed by renal biopsy;
4. Subjects with systolic blood pressure ≤ 140 mmHg and diastolic blood pressure ≤ 90 mmHg at screening;
5. If taking ACEI(Angiotensin converting enzyme inhibitors), ARB(Angiotensin receptor blocker), a stable dose within 4 weeks before screening is required;
6. Subjects who are able to follow the study protocol as judged by the investigator.

Exclusion Criteria:

1. Subjects with secondary membranous nephropathy;
2. Subjects with uncontrolled blood pressure as judged by the investigator within 3 months before screening;
3. Subjects with decreases in urine protein ≥ 50% within 6 months before screening;
4. Subjects who have received or are receiving renal replacement therapy;
5. Subjects with type 1 diabetes mellitus, or those with type 2 diabetes mellitus who are diagnosed as diabetic nephropathy by percutaneous renal biopsy;
6. Subjects who have a clear history of tuberculosis or have received anti-tuberculosis treatment;
7. Subjects with active bacterial, viral, fungal, mycobacterial, parasitic or other infections requiring systemic antibiotics or antiviral therapy;
8. Subjects with known history of severe allergic reactions to humanized monoclonal antibodies；
9. Subjects who received live vaccination, major surgery, or participated in other clinical trials within 28 days before receiving the study drug;
10. Pregnant or lactating women; women of childbearing potential who have not been sterilized do not agree to use appropriate contraceptive measures during treatment and for at least 12 months after the last dose of the study drug;
11. Subjects with serious, progressive, or uncontrolled disease that may increase risks during the participation in the study as assessed by the investigator;
12. Subjects with a history of alcoholism or drug abuse within 12 months;
13. Subjects with positive hepatitis B surface antigen; those with positive hepatitis C virus antibody; those with a history of immunodeficiency;
14. Subjects with CD4+ T lymphocyte count < 300 cells/μL;
15. Other conditions unsuitable for participation in this study determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity（DLT） | Approximately 1 years
  Adverse reactions that are certainly or possibly related to the drug being tested during the dose escalation phase.
Security: Incidence of Treatment-Emergent Adverse Events | Approximately 2 years
  Adverse event type, incidence, duration, correlation with study drug

SECONDARY OUTCOMES:
PK (Pharmacokinetics) | Approximately 1 years
  Cmax
PK (Pharmacokinetics) | Approximately 1 years
  Tmax
PK (Pharmacokinetics) | Approximately 1 years
  AUC0-last（Area Under Curve of 0-last）
Biomarkers | Approximately 1 years
  Changes in serum anti-PLA2R(Antiphospholipase A2 receptor) antibody levels relative to baseline
Immunogenicity | Approximately 1 years
  Incidence of ADA(Adenosine deaminase)
Dynamics of pharmacodynamics | Approximately 1 years
  Changes of peripheral blood CD19+B cells(B-lymphocyte antigen CD19) relative to baseline
Proportion of subjects achieving clinical remission | Approximately 2 years
  Proportion of subjects achieving clinical remission

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, He'nan
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital,College of Medicine,Zhejiang University, Hangzhou, Zhejiang
  - Peking university first hospital, Beijing
  - Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai